CLINICAL TRIAL: NCT06245681
Title: Effects of Cross-sex Hormone Treatment on Cardiac Function, Myocardial and Hepatic Fat Content, Its (Anti)-Atherogenic Implications and Effects on the Insulin System: a Pilot Study
Brief Title: Effects of Cross-sex Hormone Treatment on Cardiac Function, Myocardial and Hepatic Fat Content
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexandra Kautzky-Willer, Principal Investigator, Medical University of Vienna
Other Study IDs: 1629/2017
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Transgender women: Transgender individuals assigned male at birth undergoing estrogen and antiandrogen hormone therapy
  Interventions: Drug: gender affirming hormone therapy
- Transgender men: Transgender individuals assigned female at birth undergoing testosterone hormone therapy
  Interventions: Drug: gender affirming hormone therapy

INTERVENTIONS:
Drug: gender affirming hormone therapy — both groups are receiving gender-affirming hormone therapy; we do not compare the groups, but look at whether hormone therapy with testosterone or estrogen might have an effect on myocardial function, organ lipid content and subcutaneous to visceral fat ratio

SUMMARY:
Background: Sex hormones are believed to play an important role in the development and progression of cardiovascular disease. However, the gender gap in onset and mortality is not yet completely understood. Transsexuals undergoing hormone therapy are a promising collective for analyzing the effects of sex hormones on atherosclerosis and other cardiovascular disease. Objectives of the study: To identify gender-specific cardiovascular changes attributed to high-dose hormone therapy in male-to-female (MtF) and female-to-male(FtM) transgender using sonography and magnet resonance spectroscopy. Study design: Longitudinal cohort study. Transsexuals will undergo two 3 Tesla MRI scan sessions: 1. baseline (before hormone treatment) and 2. after 6 months of treatment. An oral glucose tolerance test (OGTT) will be performed at baseline and 6 months after treatment onset. An overall study duration of 12 months is proposed.

Materials and Methods: MRI measurements will be performed on a 3 Tesla scanner. Study population: 10 FtM, 10 male-to-female MtF transsexuals (aged 18-50), free of hormone-medication at baseline. Relevance and implications of the study: Changes in atherosclerotic risk due to hormone therapy have been studied to no definite results and so far, little is known about the effects of hormone therapy on hepatic and myocardial fatty tissue. Hence this study will provide important new data on the broad clinical aspects of sex hormones as hormone replacement therapy in particularly opposite-sex hormone therapy.

DETAILED DESCRIPTION:
Background Atherosclerosis has been shown to differ in men and women regarding disease risk, onset time and overall mortality. This gender gap is mostly attributed to sex hormones. Pre-menopausal women have less atherosclerosis risk than men of the same age; on the other hand, however, overall mortality due to cardiovascular disease is higher in women. Nonalcoholic fatty liver which is associated with liver cirrhosis and higher atherosclerotic risk due to impaired liver function is more common in men and postmenopausal women as well. Therefore, a protective effect of estrogen has been proposed. Excessive androgens on the contrary have been associated with atherogenic effects. Thus, men with high exogenous testosterone supply show higher atherosclerosis risk as do women suffering from polycystic ovary syndrome and hence hyperandrogenemia while men with an androgen deficit have an increased risk of atherosclerosis as well. Nonetheless, these findings could not be backed up by clinical intervention studies yet and further research on this gender gap is necessary. Transsexuals are usually treated with high-dose opposite-sex hormone therapy at least for one year before they undergo operations. Therefore, they are an auspicious collective to study hormone-dependent changes in atherosclerosis risk and lipid profile. Even though it has been shown that lipoproteins change during hormone therapy, leading to an increase in triglycerides and cholesterol, significant effects on atherosclerotic risk have not yet been detected. However, there is hardly any data yet available on the effect of hormone therapy on cardiovascular risk factors and morbidities as nonalcoholic fatty liver, increased fatty tissue in the myocardial cells. Effects on heart function may exist as well since elevated lipids can induce cardiac steatosis and hence diminish the diastolic heart function.

Furthermore, hormone therapy has been associated with elevated blood pressure. However, while the increased cholesterol and triglycerides may boost the risk, estrogen is believed to be a protective factor. Therefore, the effects of hormone therapy on cardiovascular disease are hard to estimate and will be further analyzed in this study. Objectives of the study

* To examine the influence of high-dose, long-term opposite-sex steroid hormone treatment on hepatic and cardiac fatty tissue and heart function in female to-male (FtM) and male-to-female (MtF) transsexuals using 3 Tesla MRS.
* To examine the influence of high-dose, long-term opposite-sex steroid hormone treatment on systolic and diastolic heart function in female to-male (FtM) and male-to-female (MtF) transsexuals using 3 Tesla MRS.
* To examine the influence of high-dose, long-term opposite-sex steroid hormone treatment on carotid-media-thickness in female to-male (FtM) and male-to-female (MtF) transsexuals using sonography.
* To examine the influence of high-dose, long-term opposite-sex steroid hormone treatment on diabetes risk and insulin sensitivity & secretion in female to-male (FtM) and male-to-female (MtF) transsexuals via the oral glucose tolerance test (OGTT) and blood sampling.

Study Design This pilot study is designed as a longitudinal mono-center study. 40 transsexual subjects (20 FtM, 20 MtF) will undergo two 3 -Tesla 1H magnet resonance spectroscopy as well as 2 sonography measurements. The first scans (baseline) will be performed before treatment, the second scans after 6 months of high-dose, long-term cross-sex hormone treatment.

Subject Section Transsexuals urging gender reassignment in a clinical setting will be enrolled in this study. 20 female-to-male (FtM) and 20 male-to-female (MtF) transsexuals will be recruited. There will be no transsexual placebo group implemented in the study because of ethical reasons. The hormone therapy they will receive is purely clinical indicated and is prescribed by a doctor not included in the study. This study does not influence either the choice nor the beginning or end of the cross-sex hormone therapy

4 METHODS AND MATERIALS Magnet Resonance Spectroscopy (MRS) MRS measurements of the heart and the liver will be done at one session at the MR Center of Excellence, Medical University of Vienna, Austria, on a 3.0-T Tim Trio System (Siemens Healthcare, Erlangen, Germany) operated with a Syngo VB15 (Siemens Healthcare) user interface as described in previous work of our group. We expect an estimated average duration of 75 minutes for:

1. 1H-magnetic resonance spectroscopy (MRS) of the liver: Measurement will be performed using a 3-T whole-body spectrometer. Localized 1H spectra will be used to quantify the hepatocellular lipid content by the series stimulated echo acquisition mode (STEAM) sequence within a volume of interest of 27 cm3.
2. 1H-magnetic resonance spectroscopy (MRS) of the heart: Retrospective ECG-gated cine true fast imaging is used to portray heart function with steady state precession (TrueFISP) sequences in two-chamber, four-chamber and short axes orientation. Left ventricular global function (end-diastolic and end-systolic volume, stroke volume, ejection fraction and myocardial mass) is computed using short axes cine series (typically 11 slices, resolution 1.4×2.1×7.0 mm3, acquisition time per segment 48ms, 25 reconstructed cardiac phases) via Argus software (Siemens Healthcare). In addition, fast low-angle shot-based retrospective ECG-gated cine phase velocity encoding sequence (velocity encoding 80 cm/s, resolution 1.7×2.1×6.0 mm3, acquisition time per segment 71ms, 20 reconstructed cardiac phases) is used to determine the E/A ratio, which is a measure of left ventricular diastolic function and is calculated as the peak velocity ratio between early (passive) filling of the ventricle during diastole (E) and late (due to atrial contraction) mitral inflow (A). Myocardial lipid measurements were performed using localized 1H-MRS based on recently introduced methods. Anatomical imaging is used to guide water suppressed pointresolved spectroscopy sequence (echo time TE 30ms, number of acquisitions (NA)=32). The volume of interest (7 cm3) is placed across the middle inter-ventricular septum. The spectral signal is acquired following ECG and navigator-based respiratory triggering using the multichannel cardiac- and spine-reception coils, both of which are provided by the system manufacturer (Siemens Healthcare). Repetition time of the sequence is given by the frequency of individual breath movement. An additional spectrum without water suppression (NA=8) is used as the internal concentration reference. The spectra are processed by the spectroscopy processing tool provided by the system manufacturer (Siemens Healthcare). The myocardial lipid content is calculated as a ratio of the sum of intensities of (CH2) (1.25 ppm) and CH3 (0.8-0.9 ppm) group resonances to the intensity of the water resonance from non-water suppressed spectra of the same volume of interest. Intensities of lipid and water resonance lines are corrected for spin-lattice (T1) and spin-spin (T2) relaxation using individual repetition time and already published T1 and T2 relaxation times of skeletal muscle at 3T.

OGTT After fasting for 8 hours' patients will be offered 75 mg of glucose solution which should be ingested within 2 minutes. Patients will receive intravenous cannulation (venflon). First HbA1C, total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, transaminases of the liver, CRP and usCRP as well as cardiovascular risk markers as adiponectine, proBNP and cell adhesion molecules (20ml) will be taken. Then blood samples will be collected 30, 60, 90, 120 and 180 minutes after glucose ingestion (20ml in total). Furthermore, a small blood sample (4ml) will be frozen and used later on for analysis of insulin, proinsulin and c-peptide if considered necessary. Finally, insulin sensitivity and secretion can be calculated from glucose, insulin and c-peptide concentration. The OGTT will be performed twice, after the initial screening and at the last screening, ergo 6 months after therapy start.

STATISTICAL AND DATA ANALYSIS Due to the explorative character of the study, a sample size calculation was not performed. The numbers of participants were generated after an interdisciplinary discussion of what is to be expected and realistic also due to the number of patients that come to the clinic and could be possible participants. Initially, the normal distribution of data will be tested using descriptive statistics.

When comparing two means from the same individual before and after 6 months if data is normally distributed a paired t-test will be conducted, if not the non-parametric Wilcoxon signed-rank test for paired samples will be applied. Comparisons of quantitative variables among groups will be performed using one-way ANOVA for parametric and Mann-Whitney test for non-parametric samples as well as at baseline as after 6 months. Correlation analysis between continuous variables will be performed by Pearson's or by Spearman's analysis, if appropriate. Levels of statistical significance will be set at p<0.05. Data will be given as mean ± SD All tests will be performed using SPSS Version 17.0, SPSS Inc., Chicago, IL.

5 ETHICAL SECTION The study will be performed in accordance with the Declaration of Helsinki (1964). There will be no placebo control in the study because a latency of more than 3 months for the start of active treatment was considered as an ethical issue and based on our experience with this subject group, will decrease compliance. All subjects will be asked for written informed consent prior to inclusion in the study and will be insured through the Department of Psychiatry in accordance with §32 of the Austrian Medicines Act. At each time subjects can decide to withdraw from the study. The investigator may remove the subjects from the trial if exclusion criteria have been met. No significant side effects are expected from the MRI measurements, sonography and OGTT.

6 HUMAN RESOURCES, STUDY SITES, COOPERATIONS The proposed research will be conducted at the Department for Endocrinology and Metabolism, Gender Medicine Unit (head Univ. Prof. Alexandra

Kautzky-Willer) and the Centre of Excellence for High-Field Magnetic Resonance (head:

Univ.-Prof. Dr.med.univ. Siegfried Trattnig, Medical University of Vienna, Austria, and the Department of Obstetrics and Gynecology, Division of Gynecologic Endocrinology and Reproductive Medicine, Unit for Gender Identity Disorder (Dr. Ulrike Kaufmann, MD). All MRI measurements will be performed on the 3T Siemens Scanner at the Centre of Excellence

7 RELEVANCE AND IMPLICATIONS OF THE STUDY To our knowledge no studies on the effects of hormone therapy in transsexuals on heart function, fat content of heart and liver have been performed yet. Studies investigating the overall cardiovascular risk changes in subjects undergoing hormone therapy could not substantiate the protective effect of estrogen or an increase of atherosclerotic events due to changes in the lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Gender Identity Disorder
* age over 18 years

Exclusion Criteria:

* age under 18 years severe neurological or internal diseases

  * steroid hormone treatment within 2 months prior to inclusion (including birth control pill, phytohormones)
  * treatment with psychotropic agents such as SSRIs
  * any implant or stainless-steel graft
  * abnormal values in routine laboratory screening or general physical examination
  * current substance abuse (determined using drug screening at the screening visit)
  * pregnancy (determined at screening visit and first MRI scan)
  * failure to comply with the study protocol or to follow the instructions of the investigating

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We included individuals solely based on gender identity
Study Population: healthy transgender persons undergoing gender-affirming hormone therapy (either testosterone or estrogen-based hormone therapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2027-10-20 (Estimated); Study Completion 2028-10-20 (Estimated)

PRIMARY OUTCOMES:
Hepatic lipid content | 6 months
  changes in the hepatic lipid content (in percent) due to long-term gender-affirming hormone therapy therapy measured by MRT
Pancreatic lipid content | 6 months
  changes in pancreatic lipid content (in percent) due to long-term gender-affirming hormone therapy therapy measured by MRT
Myocardial lipid content | 6 months
  changes in myocardial lipid content (in percent) due to long-term gender-affirming hormone therapy therapy measured by MRT
Cardiac function | 6 months
  the effect of the hormone therapy on heart function (systolic and diastolic)
Changes in insulin sensitivity via OGTT | 6 months
  changes in insulin sensitivity via OGTT
changes in insulin secretion via OGTT | 6 months
  changes in insulin secretion via OGTT

CONTACTS AND LOCATIONS:
Locations (1):
- Chiari Stoffwechselambulanz, Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Deischinger C, Slukova D, Kosi-Trebotic L, Harreiter J, Nopp S, Just I, Klepochova R, Krssak M, Trattnig S, Kaufmann U, Kautzky-Willer A. Gender-affirming hormone therapy and its impact on myocardial mass and cardiac function: a prospective magnetic resonance cohort study on transgender men and women. Eur J Endocrinol. 2025 Mar 27;192(4):429-436. doi: 10.1093/ejendo/lvaf057. PMID 40153614